CLINICAL TRIAL: NCT05348330
Title: Mid-point to Pleura Transverse Process Continuous Block Versus Thoracic Intervertebral Foramen Continuous Block, for Analgesia in Polytraumatic Patients with Multiple Rib Fractures
Brief Title: Mid-point to Pleura Transverse Process Block Versus Thoracic Intervertebral Foramen Block
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: San Salvatore Hospital of L'Aquila (Other)
Responsible Party: Principal Investigator, Emiliano Petrucci, Medical Doctor, San Salvatore Hospital of L'Aquila
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 10814/21
Record Dates: First submitted 2022-04-02; First posted 2022-04-27 (Actual); Last update posted 2024-12-03 (Actual); Status verified 2024-11

CONDITIONS: Pain, Acute; Rib Fractures; Polytrauma
Keywords: Analgesia; Local anesthetics; Myofascial block; Ultrasound guidance
MeSH Terms: conditions — Acute Pain; Rib Fractures; Multiple Trauma; Agnosia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Thoracic intervertebral foramen block (Experimental): Under ultrasound guidance the continuous thoracic intervertebral foramen block, will be provided to achieve analgesia in polytraumatic patients with rib fractures. A set for continuous peripheral nerve block will be used. The infusion rate of analgesic solution (levobupivacaine 0.25% combined with dexamethasone 16 mg) will be titrated to patient perceived pain.
  Interventions: Procedure: Thoracic intervertebral foramen block
- Mid-point to pleura transverse process block (Active Comparator): Under ultrasound guidance the continuous mid-point to pleura transverse process block, will be provided to achieve analgesia in polytraumatic patients with rib fractures. A set for continuous peripheral nerve block will be used. The infusion rate of analgesic solution (levobupivacaine 0.25% combined with dexamethasone 16 mg) will be titrated to patient perceived pain.
  Interventions: Procedure: Mid-point to pleura transverse process block

INTERVENTIONS:
Procedure: Thoracic intervertebral foramen block — Under ultrasound guidance the continuous thoracic intervertebral foramen block, will be provided to achieve analgesia in polytraumatic patients with rib fractures. A set for continuous peripheral nerve block will be used. The infusion rate of analgesic solution (levobupivacaine 0.25% combined with dexamethasone 16 mg) will be titrated to patient perceived pain. The block will be performed close, by considering the level of rib fractures.
  Arms: Thoracic intervertebral foramen block
Procedure: Mid-point to pleura transverse process block — Under ultrasound guidance the continuous mid-point to pleura transverse process block, will be provided to achieve analgesia in polytraumatic patients with rib fractures. A set for continuous peripheral nerve block will be used. The infusion rate of analgesic solution (levobupivacaine 0.25% combined with dexamethasone 16 mg) will be titrated to patient perceived pain. The block will be performed close, by considering the level of rib fractures.
  Arms: Mid-point to pleura transverse process block

SUMMARY:
The analgesic effect of continuous mid-point to pleura transverse process block compared to the analgesic effect of continuous thoracic intervertebral foramen block, in patients with multiple rib fractures.

DETAILED DESCRIPTION:
The analgesic effect of continuous mid-point to pleura transverse process block will be compared to the analgesic effect of continuous thoracic intervertebral foramen block, in patients with multiple rib fractures, by using the numeric rating scale (NRS) for pain.

ELIGIBILITY:
Inclusion Criteria:

* ribs fracture after polytrauma

Exclusion Criteria:

* pregnancy
* allergy to anesthetics
* head trauma
* history of neurological impairment (primary or secondary)
* history of cancer
* history of chronic obstructive pulmonary disease
* infections of skin close to the block site
* systemic infections

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2022-12-04 (Actual); Primary Completion 2024-10-31 (Actual); Study Completion 2024-11-28 (Actual)

PRIMARY OUTCOMES:
Pain intensity | First 72 hours from the block
  The 11-point numeric scale ranges from '0' representing one pain extreme (e.g. "no pain") to '10' representing the other pain extreme (e.g. "pain as bad as you can imagine" or "worst pain imaginable"

SECONDARY OUTCOMES:
Diaphragmatic motion | First 72 hours from the block
  The percentage of diaphragmatic thickening measured as thickness at end-inspiration-thickness at end-expiration divided by thickness at end-expiration
Arterial blood gas analysis | First 72 hours from the block
  Fraction of inspired oxygen to partial pressure of oxygen ratio
Airflow rate | First 72 hours from the block
  Patient airflow rate measured in mL/second, by using an incentive spirometer with three balls
Blood pressure | First 72 hours from the block
  Invasive blood pressure (systolic and diastolic pressure in mmHg)
Sensory block | First 72 hours from the block
  Response to the stimulus (yes or no), by using a piece of cotton, and ice in a finger of surgical glove on the patient's skin.
Request of analgesic drugs | First 72 hours from the block
  Consumption of analgesic drugs (equivalent mg of morphine)
Anesthetic spread | First 72 hours from the block
  Thoracic paravertebral space spread (yes or no), evaluated with ultrasonography
Complication | First 72 hours from the block
  Number of pneumothorax, hemothorax, hematoma, pain, infection, and neurological impairment by the block

CONTACTS AND LOCATIONS:
Overall Officials: Emiliano Petrucci, MD, Principal Investigator — San Salvatore Acadec Hospital of L'Aquila (Italy)
Locations (1):
- Emiliano, L’Aquila, L'Aquila, Italy

IPD SHARING:
Plan to Share IPD: No